CLINICAL TRIAL: NCT01153633
Title: Pilot, Randomised, Double-blind, Controlled Clinical Trial on the Combined Efficacy of Prontosan Wound Irrigation Solution and Prontosan Wound Gel in the Reduction in Size and Change in Bioburden of Hard-to-heal Venous Leg Ulcers
Brief Title: Trial on the Efficacy of Prontosan Wound Irrigation Solution and Prontosan Wound Gel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: B. Braun Ltd. Centre of Excellence Infection Control (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OPM-G-H 0901
Record Dates: First submitted 2010-06-28; First posted 2010-06-30 (Estimated); Results first posted 2014-04-01 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prontosan Wound Solution and Gel (Active Comparator): Cleansing the wound bed, a sterile gauze dressing impregnated with the Prontosan® or saline solution, removed after 15 minutes; wound will be sparingly covered with Prontosan® Wound Gel or inactive gel. Secondary dressing to be a semi occlusive dressing. Secure the dressing to the wound with tubifast and short stretch compression system Dressings will be changed and the treatment procedure will be repeated every 3 days (+/- 1 day)
  Interventions: Device: Prontosan Wound Irrigation Solution and Prontosan Wound Gel
- Normal Saline and Placebo Gel (Placebo Comparator): Cleansing the wound bed, a sterile gauze dressing impregnated with the Prontosan® or saline solution, removed after 15 minutes; wound will be sparingly covered with Prontosan® Wound Gel or inactive gel. Secondary dressing to be a semi occlusive dressing. Secure the dressing to the wound with tubifast and short stretch compression system Dressings will be changed and the treatment procedure will be repeated every 3 days (+/- 1 day)
  Interventions: Device: Normal Saline and Placebo Gel

INTERVENTIONS:
Device: Prontosan Wound Irrigation Solution and Prontosan Wound Gel — The treatment procedures (after a 1 week run-in) include:
  * Cleansing the wound bed, at dressing change, with Prontosan® Wound Irrigation Solution or saline solution; a sterile gauze dressing impregnated with the Prontosan® or saline solution, depending on randomisation, will be placed on the wound in the form of a moist compress and removed after 15 minutes; the wound will be sparingly covered with Prontosan® Wound Gel or inactive gel, depending on randomisation
  * Secondary dressing to be a semi occlusive dressing
  * Secure the dressing to the wound with tubifast and short stretch compression system Dressings will be changed and the treatment procedure will be repeated every 3 days (+/- 1 day) when clinical, microbiological, planimetry and photographic assessments will be made. The randomised solution will also be used for removal of the dressing from the wound at the start of dressing change.
  Arms: Prontosan Wound Solution and Gel
Device: Normal Saline and Placebo Gel — The treatment procedures (after a 1 week run-in) include:
  * Cleansing the wound bed, at dressing change, with Prontosan® Wound Irrigation Solution or saline solution; a sterile gauze dressing impregnated with the Prontosan® or saline solution, depending on randomisation, will be placed on the wound in the form of a moist compress and removed after 15 minutes; the wound will be sparingly covered with Prontosan® Wound Gel or inactive gel, depending on randomisation
  * Secondary dressing to be a semi occlusive dressing
  * Secure the dressing to the wound with tubifast and short stretch compression system
  Dressings will be changed and the treatment procedure will be repeated every 3 days (+/- 1 day) when clinical, microbiological, planimetry and photographic assessments will be made. The randomised solution will also be used for removal of the dressing from the wound at the start of dressing change.
  Arms: Normal Saline and Placebo Gel

SUMMARY:
The primary objective of the study is to evaluate the efficacy of Prontosan® Wound Irrigation Solution and Prontosan® Wound Gel in the treatment of hard-to heal venous leg ulcers compared to control saline irrigation solution and inactive gel by showing a reduction in size over a 12 week period.

DETAILED DESCRIPTION:
SUMMARY

Sponsor: B. BRAUN Medical AG

Trade name: Prontosan® Wound Irrigation Solution Prontosan® Wound Gel

Active substance: Polihexanide (0.1%) Betaine (0.1%)

Study Duration (per patient):

13 weeks, including the 1 week run in period

Primary Objective:

To evaluate the efficacy of the combination of Prontosan® Wound Irrigation Solution and Prontosan® Wound Gel in the reduction of wound size of hard-to-heal venous leg ulcers compared to control saline irrigation solution and inactive gel.

Secondary Objectives:

To assess the change in bio-burden (assessment of organisms present) and to determine local tolerance as well as reduction in pain and to monitor exudate control.

Methodology:

A pilot randomised, double-blind, controlled clinical trial at a single centre

Planned number of patients:

A sample size of N= 15 evaluable patients was estimated for each treatment group (group "A" and "B"). Adding a dropout rate of approx. 25% results in a total number of patients for both treatment groups of N=38.

Study Visits:

Visit 0 (-1 week) - Screening Visit 1 ( Week 0) - Treatment and assessment visit Visit 2 (Week 1, day 7 +/- 1 day) - Treatment and assessment visit Visit 3 (Week 2, day14 +/- 1 day) - Treatment and assessment visit Visit 4 (Week 4, day 28 +/- 2 days) - Treatment and assessment visit Visit 5 (Week 8, day 56 +/- 2 days) - Treatment and assessment visit Visit 6 (Week 12, day 84 +/- 2 days) - End of study following 12 weeks of treatment or at healing whichever is soonest

The number of additional visits will be recorded in the Case Report Forms.

Treatment efficacy assessment:

Clinical signs and symptoms will be compared between the two randomised groups with microbiological analysis and, computer planimetry assessments of ulcer size, using Visitrak™ (Smith & Nephew), and digital photography at entry to the study, at each planned study visit and at healing or 12 weeks, whichever is soonest.

Tolerance assessment:

The tolerability of study treatment will be evaluation based on the intensity and the course of adverse events (undesired concomitant effects, both subjectively perceived symptoms and objectively detected signs of disease). Tolerance assessments will take place from visit 2 onwards

Assessment methods:

1. Assessment of clinical signs and symptoms, in particular related to development of infection:

   * reduction of slough and necrotic tissue
   * control of exudate
   * presence of granulation tissue
   * reduction of inflammatory signs (surrounding skin)
   * pain
2. Ulcer computerised planimetry using Visitrak™
3. Microbiological analysis for bioburden (the bioburden within an ulcer relates to a microbiological qualitative and quantitative assessment of organisms present) assessed by wound swab or biopsy
4. Serial photography with blinded assessment of progress using linear analogue scale

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged > 18 who are able to give informed consent
* Patients with a chronic venous leg ulcer at any location below the knee joint (CVI grade C6 according to CEAP classification = trophic lesions and open ulcer)
* Venous leg ulcer present for ≥4 weeks
* Surface area of the target ulcer ≥2cm2 and <100cm2 with the largest length not being >10cm
* ABPI ≥ 0.7

Exclusion Criteria:

* Age below 18 years
* Females of child bearing potential who are not willing to use a method of highly effective contraception during the entire study
* Pregnant or breast feeding women
* Signs and symptoms of clinical infection, or current use of antiseptics or antibiotics
* Involvement in other trials within the past 1 month
* Sensitivity to any of the components of Prontosan® or dressing material
* Intolerance to compression therapy
* Active osteomyelitis in the ulceration area
* Active rheumatoid or collagen disease of blood vessels treated with corticosteroids
* Chronic diseases that could impact the course of the study (malicious cancer, TB, AIDS, mental illnesses)
* Plasma protein below 4 g/dl
* Anaemia: haemoglobin below 10 g/dl
* Poorly controlled Diabetes (HBA1C > 12%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Harding, MD, Principal Investigator — Cardiff University, Department of Wound Healing
Locations (1):
- Cardiff University, Department of Wound Healing, Cardiff, Wales, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Prontosan Wound Solution and Gel: Polihexanide (0.1%), Betaine (0,1%), Purifed water
- Normal Saline and Placebo Gel: Sodium Chloride 0.9% Solution Inactive Hydrogel, Hydroxyethylcellulose, Glycerol, purified water, exipients
Period: Overall Study
Arm/Group | Prontosan Wound Solution and Gel | Normal Saline and Placebo Gel
Started | 17 | 17
Completed | 13 | 13
Not Completed | 4 | 4
Not completed — Protocol Violation | 1 | 1
Not completed — Therapeutic failure | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Normal Saline and Placebo Gel: Sodium Choride 0.9% Solution, Neutral Gel without Polihexanide, without Betaine
- Total: Total of all reporting groups
Arm/Group | Prontosan Wound Solution and Gel | Normal Saline and Placebo Gel | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.1 (9.6) | 73.1 (10.7) | 71.6 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 19
  Male | 5 | 10 | 15
Region of Enrollment [Number; unit: participants]
  United Kingdom | 17 | 17 | 34
Duration of leg ulceration [Median (Full Range); unit: months] | 36 [5 to 360] | 84 [3 to 84] | 54 [3 to 384]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change of Wound Size From Baseline to Last Visit
Time Frame: 12 Weeks
Population: Per protocol set
Measure: Least Squares Mean (Standard Error); unit: percentage change in wound size (cm2)
Groups:
- Prontosan Wound Irrigation Solution and Gel: Polihexanide 0.1%, Betaine 01.%, purified water, exipients
- Normal Saline and Inactive Gel: Sodium Chloride 0.9% Solution Inactive Hydrogel, Hydroxyethylcellulose, Glycerol, purified water, exipients
Arm/Group | Prontosan Wound Irrigation Solution and Gel | Normal Saline and Inactive Gel
Number analyzed (Participants) | 17 | 15
percentage change in wound size (cm2) | -64.98 (12.32) | -42.78 (13.13)
Statistical Analysis 1: Comparison: Prontosan Wound Irrigation Solution and Gel vs Normal Saline and Inactive Gel; Test type: Superiority or Other; p = 0.2317, F-test — F-test (2-sided), ANCOVA with baseline target ulcer size as covariate

2. Secondary Outcome: Number of Different Microganisms at V6/EoS
Time Frame: 12 Weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: Number of microgasism species
Groups:
- Prontosan Wound Solution and Gel: Polihexanide 0.1%, Betaine 0.1%, purified water, exipients
Arm/Group | Prontosan Wound Solution and Gel | Normal Saline and Placebo Gel
Number analyzed (Participants) | 17 | 15
Number of microgasism species | 0.8 (0.9) | 1.0 (0.8)

3. Secondary Outcome: Pain
Description: Absolute change (mm VAS) from baseline to V6/EoS. Pain intensity assessed by patient. At each study visit the patients assessed their pain intensity using a 100 mm Visual Analogue Scale (VAS). Thereby 0 mm represented 'no pain' and 100 mm 'worst possible pain'.
Time Frame: 12 Weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Prontosan Wound Solution and Gel | Normal Saline and Placebo Gel
Number analyzed (Participants) | 17 | 15
mm | -8.9 (20.4) | -12.8 (26.0)

4. Secondary Outcome: Condition of Wound Bed
Description: Sum of granulation and epithelium (% of wound bed), absolute change from baseline to V6/EoS
Time Frame: 12 Weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: percentage of of wound bed
Arm/Group | Prontosan Wound Solution and Gel | Normal Saline and Placebo Gel
Number analyzed (Participants) | 17 | 15
percentage of of wound bed | 7.1 (38.9) | -1.5 (52.0)

5. Primary Outcome: Healing of Target Ulcer atV6/EOS
Description: Number of ulcers healed at V6/EOS
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Number; unit: ulcers
Arm/Group | Prontosan Wound Solution and Gel | Normal Saline and Placebo Gel
Number analyzed (Participants) | 17 | 15
ulcers | 8 | 5
Statistical Analysis 1: Comparison: Prontosan Wound Solution and Gel vs Normal Saline and Placebo Gel; Test type: Superiority or Other; p = 0.4905, Fisher Exact

6. Primary Outcome: Absolute Change of Target Ulcer From Baseline to Last Visit
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Least Squares Mean (Standard Error); unit: square centimeters
Arm/Group | Prontosan Wound Solution and Gel | Normal Saline and Placebo Gel
Number analyzed (Participants) | 17 | 15
square centimeters | -3.00 (1.45) | -3.01 (1.54)
Statistical Analysis 1: Comparison: Prontosan Wound Solution and Gel vs Normal Saline and Placebo Gel; Test type: Superiority or Other; p = 0.9945, F-test — F-test (2-sided), ANCOVA with baseline target ulcer size as covariate

ADVERSE EVENTS:
Arm/Group | Prontosan Wound Solution and Gel | Normal Saline and Placebo Gel
Serious Adverse Events (participants affected / at risk) | 0/17 | 1/17
Other Adverse Events (participants affected / at risk) | 15/17 | 15/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prontosan Wound Solution and Gel (N=17) | Normal Saline and Placebo Gel (N=17)
Chest Pain (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prontosan Wound Solution and Gel (N=17) | Normal Saline and Placebo Gel (N=17)
Celulitis (Infections and infestations) | 1 (1) | 1 (1)
Infected skin ulcer (Infections and infestations) | 5 (7) | 4 (4)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 5 (6) | 4 (5)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Skin maceration (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (2) | 3 (6)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 7 (11) | 6 (6)
Venous ulcer pain (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Skin chapped (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Most likely the non-statistical significant results are due to the small sample size. No sample size calculation and statistical analysis was planned a priori because it was a pilot study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No